CLINICAL TRIAL: NCT00551629
Title: Safety, Tolerability, and Immunogenicity of Four Different Formulations of a Liquid Hexavalent Combination Vaccine, HR5I (Haemophilus Influenzae Type b Conjugate, Recombinant Hepatitis B Surface Antigen, Diphtheria Toxoid, Tetanus Toxoid, 5-Component Acellular Pertussis Vaccine, and Inactivated Poliovirus Type 1, 2, and 3), When Administered to Healthy Hepatitis B Vaccine-Naïve Infants at 2, 3, 4, and 12 to 14 Months of Age
Brief Title: A Study to Test the Safety and Effectiveness of an Investigational Vaccine in Infants (V419-002)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V419-002; 2007_580 (Other: Merck Registration Number)
Record Dates: First submitted 2007-10-29; First posted 2007-10-31 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Bacterial Infections; Virus Diseases
MeSH Terms: conditions — Bacterial Infections; Virus Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- AR51 (12, 10) (Experimental): Participants were vaccinated with 0.5 ml of AR51 (12, 10) formulation via intramuscular injection as a primary series at 2, 3, and 4 months of age, and as a booster at 12 to 14 months of age.
  Interventions: Biological: AR51 (12, 10)
- PR51 (3, 10) (Experimental): Participants were vaccinated with 0.5 ml of PR51 (3, 10) formulation via intramuscular injection as a primary series at 2, 3, and 4 months of age, and as a booster at 12 to 14 months of age.
  Interventions: Biological: PR51 (3, 10)
- PR51 (6, 10) (Experimental): Participants were vaccinated with 0.5 ml of PR51 (6, 10) formulation via intramuscular injection as a primary series at 2, 3, and 4 months of age, and as a booster at 12 to 14 months of age.
  Interventions: Biological: PR51 (6, 10)
- PR51 (6, 15) (Experimental): Participants were vaccinated with 0.5 ml of PR51 (6, 15) formulation via intramuscular injection as a primary series at 2, 3, and 4 months of age, and as a booster at 12 to 14 months of age.
  Interventions: Biological: PR51 (6, 15)

INTERVENTIONS:
Biological: AR51 (12, 10) — vaccine formulation containing 12 mcg of PRP-T and 10 mcg of HBsAg
  Arms: AR51 (12, 10)
Biological: PR51 (3, 10) — vaccine formulation containing 3 mcg of PRP-OMPC and 10 mcg of HBsAg
  Arms: PR51 (3, 10)
Biological: PR51 (6, 10) — vaccine formulation containing 6 mcg of PRP-OMPC and 10 mcg of HBsAg
  Arms: PR51 (6, 10)
Biological: PR51 (6, 15) — vaccine formulation containing 6 mcg of PRP-OMPC and 15 mcg of HBsAg
  Arms: PR51 (6, 15)

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and immunogenicity of 4 different formulations of the HR5I vaccine (Haemophilus influenzae type b conjugate, recombinant hepatitis B surface antigen, diphtheria, tetanus, 5-component acellular pertussis, and inactivated poliovirus Types 1, 2, and 3). The primary hypothesis is that at least 1 of the 4 formulations of HR5I administered as a primary series at 2, 3, and 4 months of age will be acceptable (similar to targeted rates) with respect to Postdose 3 antibody responses to all antigens.

DETAILED DESCRIPTION:
Participants will be randomized into 4 arms:

AR51 (12, 10): arm receiving vaccine formulation containing 12 mcg of polyribosylribitol phosphate (PRP) conjugates to tetanus toxoid (PRP-T) and 10 mcg of Hepatitis B surface antigen (HBsAg)

PR51 (3, 10): arm receiving vaccine formulation containing 3 mcg of PRP conjugated to the outer membrane protein complex of Neisseria meningitides (PRP-OMPC) and 10 mcg of HBsAg

PR51 (6, 10): arm receiving vaccine formulation containing 6 mcg of PRP-OMPC and 10 mcg of HBsAg

PR51 (6, 15): arm receiving vaccine formulation containing 6 mcg of PRP-OMPC and 15 mcg of HBsAg

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants 2 months of age who have not received prior vaccinations for Haemophilus influenzae type b (Hib), hepatitis B, Diptheria/Pertussis/Tetanus (DPT), or Polio

Exclusion Criteria :

* Documented HIV infection (child or mother)
* Documented HBsAg-seropositivity (child or mother)
* History of invasive Hib disease, hepatitis B, diphtheria, tetanus, pertussis, or poliovirus infection
* History of seizure disorder, developmental delay, or any other neurologic disorder
* Underlying medical conditions such as inborn errors of metabolism, failure to thrive, or any major congenital abnormalities requiring surgery
* Prior or anticipated receipt of immune globulin, blood, or blood products
* Known hypersensitivity to any component of the investigational vaccines being administered in this protocol
* Any history or condition that would exclude the child from receiving any vaccine administered under this protocol
* Any condition that, in the opinion of the investigator, may interfere with the evaluation of the study objectives

Ages: 6 Weeks to 9 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 708 (Actual)
Dates: Start 2001-05; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with level of anti-PRP antibodies >1.0 μg/mL at the Postdose 3 time point | At 5 months of age (1 month after 3rd vaccination)
Percentage of participants with level of anti-HBsAg antibodies ≥10 mIU/L at the Postdose 3 time point | At 5 months of age (1 month after 3rd vaccination)
Percentage of participants with a ≥4-fold rise in levels of antibodies to pertussis antigens (toxoid [PTxd], Filamentous Hemagglutinin [FHA], Fimbria 2 & Fimbria 3 [FIM], and Pertactin [PRN]) at the Postdose 3 time point | At 5 months of age (1 month after 3rd vaccination)
Percentage of participants with level of anti-diphtheria antibodies ≥0.01 IU/mL at the Postdose 3 time point | At 5 months of age (1 month after 3rd vaccination)
Percentage of participants with level of anti-tetanus antibodies ≥0.01 IU/mL at the Postdose 3 time point | At 5 months of age (1 month after 3rd vaccination)
Percentage of participants with neutralizing anti-poliovirus antibodies (Types 1, 2, and 3) at ≥1:8 dilution at the Postdose 3 time point | At 5 months of age (1 month after 3rd vaccination)

SECONDARY OUTCOMES:
Number of participants with at least 1 adverse event (AE) | From 1st vaccination up to 14 days following last vaccination (up to 14.5 months)
Number of participants who discontinued study treatment due to an AE | From 1st vaccination up to 14 days following last vaccination (up to 14.5 months)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Halperin SA, Tapiero B, Diaz-Mitoma F, Law BJ, Hoffenbach A, Zappacosta PS, Radley D, McCarson BJ, Martin JC, Brackett LE, Boslego JW, Hesley TM, Bhuyan PK, Silber JL. Safety and immunogenicity of a hexavalent diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine at 2, 3, 4, and 12-14 months of age. Vaccine. 2009 Apr 28;27(19):2540-7. doi: 10.1016/j.vaccine.2008.11.115. Epub 2009 Jan 3. PMID 19124057